CLINICAL TRIAL: NCT07123649
Title: Individualizing Approaches to Surveillance Mammography in Older Breast Cancer Survivors - The I-MAMMO Study
Acronym: I-MAMMO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-122; 1R01AG089237-01 (NIH)
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Cancer Survivor; Breast Cancer Survivorship
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized at the clinician level in a 1:1 fashion, stratified by site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shared-Decision Making Toolkit (Experimental): Enrolled participants will complete:
  * Year 1 standard of care visit with clinician followed by post-visit survey
  * Optional semi-structured interview with study staff
  * Year 2 standard of care visit with clinician followed by post-visit survey
  * Optional semi-structured interview with study staff
  * End of study survey
  Interventions: Behavioral: Shared Decision-Making Toolkit
- Usual Care (No Intervention): Enrolled participants will continue with standard care practices without the SDM toolkit and will complete:
  * Year 1 standard of care visit with clinician followed by post-visit survey
  * Year 2 standard of care visit with clinician followed by post-visit survey
  * Optional semi-structured interview with study staff

INTERVENTIONS:
Behavioral: Shared Decision-Making Toolkit — The SDM toolkit is designed to support discussions on the continuation of surveillance mammography. It provides evidence-based guidelines, communication strategies, and education materials to aid in personalized decision-making.
  Other Names: SDM Toolkit
  Arms: Shared-Decision Making Toolkit

SUMMARY:
This study evaluates the effectiveness of a Shared Decision-Making (SDM) toolkit designed to support older breast cancer survivors aged 80 and above in making informed decisions about continuing surveillance mammography.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of a Shared Decision-Making (SDM) toolkit designed to support older breast cancer survivors aged 80 and above in making informed decisions about continuing surveillance mammography.

A participant will be placed into one of two groups: Group A: Usual Care vs. Group B: SDM Toolkit according to the randomized placement of the assigned study clinician.

Study procedures include questionnaires and option interviews with study staff.

Participation in this research study is expected to last about 2 years.

It is expected about 52 clinicians and 312 participants will take part in this research study.

The National Institute on Aging is providing funding for this research study

ELIGIBILITY:
Participant Inclusion Criteria:

* Women aged ≥ 80 years at the time of registration
* History of stage 0-III breast cancer (Of note: ductal carcinoma in situ [DCIS], pleomorphic lobular carcinoma in situ [because it is typically treated like DCIS], or invasive breast cancer of any subtype are all eligible)
* No history of a recurrent breast cancer (i.e., a breast cancer that is deemed metastatic or a locoregional recurrence of a prior cancer per clinician judgement rather than a new primary breast cancer). If a person has been diagnosed with multiple distinct breast cancers over time (e.g., history of left and right breast cancer), they are eligible as long as they meet other requirements for time since surgery, etc.
* Has at least one intact breast
* Has had mammogram screening/surveillance within the last 24 months

  -≥ 12 months since most recent breast surgery to affected breast (e.g., breast reduction surgery on an unaffected breast within 12 months is ok)
* No active cancer-directed therapy other than hormonal therapy and/or CDK 4/6 inhibitor therapy
* Ability and willingness to take surveys
* Receiving at least some of their oncology follow-up care at a participating site
* Most recent mammogram report for the potential participant did not recommend additional diagnostic work-up or close interval follow-up imaging

  * If a patient required diagnostic breast testing in the past or at the time of the most recent mammogram AND the results were resolved to benign findings with no additional diagnostics recommended, they are eligible.
  * If a patient's most recent mammogram result isn't yet available at the time of approach or study consent, the patient is eligible to proceed with consent and enrollment. If this mammogram then abnormal or requires additional imaging, that patient will not be included in the study analyses or surveys. This patient will be replaced.

Participant Exclusion Criteria:

* Inability to provide informed consent
* Assigned male sex at birth
* Breast or recent imaging findings requiring diagnostic testing at baseline
* Prior discontinuation of mammography by electronic medical record (EMR) review or patient report
* Prior atypical ductal hyperplasia (ADH) or non-pleomorphic LCIS only
* Psychiatric illness situations that would limit compliance with study requirements
* Those with metastatic breast cancer
* Those in hospice care
* Those whose clinician is not willing to participate
* Pregnant women, young patients, and those in prison will not be eligible for enrollment given the study design and aims supporting study in a different population focused on older adults

Clinician Inclusion Criteria:

* Must be an active clinician (MD, NP, or PA) at a participating institution
* Sees at least one breast-cancer survivor aged ≥ 80
* Clinician must be able to read, speak, and write in English

Min Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Mammography Rate | Assessed at 2 years post-enrollment.
  Mammography Rate is defined as the proportion of participants that undergo mammography by 2 years post-enrollment.

SECONDARY OUTCOMES:
Mammography Count | Assessed at 2 years post-enrollment.
  Mammography Count is defined as the count of all mammograms each participant underwent during study follow-up.
Participant Knowledge Score | Annually through 2 years of follow-up post-enrollment.
  Participant Knowledge Score will be defined as the proportion of correct knowledge questions (range: 0 to 1).
Participant Decisional Quality Score | Annually through 2 years of follow-up post-enrollment.
  Participant Decisional Quality Score will be defined as the sum of response scores (range of 0-4), with each individual response scored 0 or 1. Higher scores indicate higher decisional quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu